CLINICAL TRIAL: NCT00893555
Title: Pharmacologic Optimization of Voriconazole - a Prospective Clustered Group-randomized Cross-over Trial of Therapeutic Drug Monitoring
Brief Title: Pharmacologic Optimization of Voriconazole
Acronym: VORI911
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jan-Willem C Alffenaar (Other)
Collaborators: University Medical Center Nijmegen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amsterdam UMC, location VUmc (Other); Leiden University Medical Center (Other); UMC Utrecht (Other); Erasmus Medical Center (Other); St. Antonius Hospital (Other); Meander Medical Center (Other); Haga Hospital (Other); Klinikum Oldenburg gGmbH (Other)
Responsible Party: Sponsor-Investigator, Jan-Willem C Alffenaar, PhD PharmD, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VORI911
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Invasive Fungal Infection; Hematological Malignancy
Keywords: Invasive fungal infection; hematological malignancy; voriconazole; therapeutic drug monitoring
MeSH Terms: conditions — Invasive Fungal Infections; Hematologic Neoplasms | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): Voriconazole dosing based on SPC
  Interventions: Drug: voriconazole (dosing according to the SPC)
- TDM (Experimental): Voriconazole serum concentration based dosing
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — TDM (through level of 2-5mg/L).
  Other Names: Vfend
  Arms: TDM
Drug: voriconazole (dosing according to the SPC) — No serum concentrations are determined
  Other Names: Vfend
  Arms: control

SUMMARY:
The objective of this study proposal is to determine whether pharmacologic optimization of voriconazole by means of therapeutic drug monitoring (TDM) results in improved patient outcomes (efficacy and safety) and is more cost-effective compared to the current standard of care.

DETAILED DESCRIPTION:
Patients with haematological malignancies and chemotherapy-induced prolonged neutropenia are at risk for severe bacterial and fungal infections. These opportunistic infections can result in prolonged hospital stay, increases costs and greater mortality. Voriconazole has now been recommended as the first line agent for invasive pulmonary aspergillosis. Retrospective observational studies of voriconazole serum concentration suggest that serum concentration correlate with toxicity and clinical response. These observations were however made in small series of patients and data were collected retrospectively. These inherent methodological flaws make it impossible to draw definite conclusions about the effect of voriconazole serum level monitoring on the outcome of IA, and therefore considered insufficient proof to recommend voriconazole concentration determination in blood as standard of care. The impact that so called serum concentration guided dosing of voriconazole will have on treatment success can only be evaluated through a prospective randomized clinical trial.

For this purpose, we designed a prospective stratified cluster randomized cross-over trial of therapeutic drug monitoring in patients with haematological disease who have developed IA. The order of periods (TDM or standard of care, each 12 months) will be randomized per centre. During the TDM episode, the voriconazole dosage will be adjusted to achieve trough blood concentrations in a predefined window of 2-5 mg/L. A sample size of n=192 is needed to detect a 20% absolute reduction in the number of treatment failures (40% to 20 %) compared to control.

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 years of age
* have received chemotherapy for haematological malignancies or have received a hematopoietic stem cell transplant
* proven, probable or possible invasive fungal disease according to the EORTC/MSG criteria
* treatment with voriconazole

Exclusion Criteria:

* allergic to voriconazole or its excipients
* age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-04; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The primary clinical endpoint will be a global response consisting of a combined endpoint of toxicity and response to therapy (clinical, microbiologic and radiologic responses) 28 days after starting treatment with voriconazole. | 28 days

SECONDARY OUTCOMES:
Overall mortality | 7 and 28 days; 12 weeks
% of serum concentrations within 2-5mg/L | 7 and 28 days; 12 weeks
% switched to salvage therapy or measured concentration level in control arm | 7 and 28 days; 12 weeks
Side effects | 7 and 28 days; 12 weeks
Time to global response | 7 and 28 days; 12 weeks
Cost-effectiveness of TDM | 7 and 28 days; 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J GW Kosterink, PharmD, PhD, Study Chair — University Medical Center Groningen; J WC Alffenaar, PharmD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Klomp SD, Veringa A, Alffenaar JC, de Boer MGJ, Span LFR, Guchelaar HJ, Swen JJ. Inflammation altered correlation between CYP2C19 genotype and CYP2C19 activity in patients receiving voriconazole. Clin Transl Sci. 2024 Jul;17(7):e13887. doi: 10.1111/cts.13887. PMID 39010708
- [Derived] Veringa A, Bruggemann RJ, Span LFR, Biemond BJ, de Boer MGJ, van den Heuvel ER, Klein SK, Kraemer D, Minnema MC, Prakken NHJ, Rijnders BJA, Swen JJ, Verweij PE, Wondergem MJ, Ypma PF, Blijlevens N, Kosterink JGW, van der Werf TS, Alffenaar JC; Voriconazole ZonMw Study Group. Therapeutic drug monitoring-guided treatment versus standard dosing of voriconazole for invasive aspergillosis in haematological patients: a multicentre, prospective, cluster randomised, crossover clinical trial. Int J Antimicrob Agents. 2023 Feb;61(2):106711. doi: 10.1016/j.ijantimicag.2023.106711. Epub 2023 Jan 13. PMID 36642232